CLINICAL TRIAL: NCT03415789
Title: Quantification of Intraventricular Stasis and Thromboembolic Risk With New Imaging Methods in Patients With Non Ischemic Dilated Myocardiopathy
Brief Title: Intraventricular Stasis in Non Ischemic Dilated Myocardiopathy
Acronym: ISBIDCM
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Javier Bermejo Thomas, Head of Cardiac Imaging. Principal Investigator., Hospital General Universitario Gregorio Marañon
Other Study IDs: FIBHGM-ISBIDCM
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Dilated Cardiomyopathy; Thrombosis; Stroke
Keywords: Non ischemic dilated cardiomyopathy; Cardiac thrombosis; Silent brain infarct; Fluid dynamics; Intracardiac blood flow; Echocardiography
MeSH Terms: conditions — Cardiomyopathy, Dilated; Thrombosis; Stroke | interventions — Blood Coagulation Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 80 patients non ischemic DCM: A cohort of 80 patients with nonischemic dilated cardiomyopathy in sinus rhythm with left ventricle ejection fraction (EF) less than 45%.
  In the first 24 hours after enrollment a coagulation blood test, an electrocardiogram, a Doppler echocardiogram exam and a clinical examination (including neuropsiquiatric evaluation) will be performed.
  A cardiac magnetic resonance and a brain magnetic resonance will be performed within 10 days after the enrollment.
  Interventions: Diagnostic Test: Doppler echocardiogram exam; Diagnostic Test: Cardiac Magnetic Resonance; Diagnostic Test: Brain Magnetic Resonance; Diagnostic Test: Coagulation blood test

INTERVENTIONS:
Diagnostic Test: Doppler echocardiogram exam — A complete echocardiographic study will be performed at enrollment. The echocardiographic images will be acquired as clinically recommended. The protocol will include the acquisition of 1) 2D images in parasternal axis long and short axis; 2) 2D and Doppler tissue images in the apical planes of 4, 2 and 3 chambers; 3) Pulsed, continuous and color Doppler M (DCMM) of transmitral LV flow and LV ejection; 4) 3-Chamber apical plane with and without color Doppler; and 5) 3D LV images. DCMM images will be obtained from the apical window using 4 and 5 chamber planes. Blood flow velocity will be obtained using Color and Gray mode in the 3 chamber view during 5-10 beats in apnea.
Diagnostic Test: Cardiac Magnetic Resonance — A cardiac MR will be acquired within 10 days after the enrollment. The protocol includes the following sequences: cine mode of short axis from LV base to apex and 2-3-4 chambers. 3D sequence of late enhancement of inversion-recovery. Images will be acquired after 3 min and 10 min of the administration of a total of 0.2 mmol / kg of Prohance®. Intraventricular thrombosis will be monitored. Phase contrast sequences in three orthogonal planes will be acquired. Morphological parameters of LV function (LVEF), contractility ("Wall Motion Score ") and sphericity index will be measured.
Diagnostic Test: Brain Magnetic Resonance — A brain MR will be acquired within 10 days after the enrollment. Axial, sagittal and coronal spin echo sequence in T1, axial images in diffusion sequences (DWI), enhanced spin echo T2 and FLAIR (fluid-attenuated inversion recovery) sequences shall be obtained. A cerebral infarction will be positive when finding the presence of a focal lesion of> 3 mm in diameter that meets one of these three characteristics: (1) high signal on isotropic DWI images and low signal on the apparent coefficient map Broadcast (ADC). (2) Cavitary lesion hyperintense on T2, with no signal (or low) in the FLAIR sequence. (3) Hyperintense lesion T2 / T1 hypointense with prior distribution defect known or new in a follow-up study.
Diagnostic Test: Coagulation blood test — 5 ml of peripheral blood will be obtained for assessment of prothrombotic markers at enrollment.

SUMMARY:
This study is designed to quantify the ventricular stasis in patients with non-ischemic dilated cardiomyopathy by post-processing of 2D color Doppler echocardiography images in order to establish the relationship between quantitative variables of intraventricular stasis and the prevalence of silent embolic events and/or intraventricular mural thrombosis determined by magnetic resonance.

DETAILED DESCRIPTION:
In patients with left ventricular dysfunction, intraventricular mural thrombosis is a recognized risk factor for cardioembolic events. The flow stasis accompanying ventricular remodeling and myocardial dysfunction could favor the formation of small intracavitary thrombi between LV trabeculae, small enough not be detected by conventional imaging techniques. Computational post-processing techniques allow a robust and complete characterization of numerous aspects of fluid dynamics within the heart using the flow field obtained by Echo or MRI imaging, and it is possible to quantify the stasis and washing of blood in the left ventricular cavity.

A cross-sectional study in 80 patients with non-ischemic DCM in sinus rhythm is proposed in which an echocardiogram, cardiac and cerebral MRI will be performed. Our objective is to quantify the ventricular stasis by post-processing of 2D color Doppler echocardiography images in order to establish the relationship between quantifiable intraventricular stasis variables and the prevalence of silent and embolic events and intracavitary thrombosis determined by magnetic resonance (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonischemic dilated cardiomyopathy.
* Sinus rhythm.
* LV ejection fraction (EF) less than 45%.
* Signature of informed consent for the study.

Exclusion Criteria:

* Implantable defibrillation or stimulation devices not compatible with MRI.
* Hemodynamically significant primary valvular disease or cardiac valve prosthesis.
* Claustrophobia.
* Documented history of paroxysmal or persistent atrial fibrillation (AF).
* Previous carotid disease diagnosed with stenosis greater than 50%.
* Complete oral anticoagulation prior to inclusion in the study or indication of anticoagulation.
* Known prothrombotic states (active oncological pathology, alteration of the coagulation cascade).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients with diagnosis of non-ischemic dilated cardiomyopathy under follow-up in the Cardiology Department of Gregorio Marañón General University Hospital, Madrid, who meet all of the inclusion criteria and none of the exclusion criteria will be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Prevalence of the combined binary variable consisting of left ventricular mural thrombosis or silent brain infarct detected by magnetic resonance imaging | Within 10 days after enrollment
  Quantification of the prevalence of the combined binary variable consisting of one of the following: ventricular thrombosis assessed by cardiac magnetic resonance or silent brain infarct detected by brain magnetic resonance.

SECONDARY OUTCOMES:
Left ventricle mural thrombosis assessed by cardiac magnetic resonance imaging | Within 10 days after enrollment
  Left ventricle mural thrombosis will be assessed by contrast cardiac MRI. Early after gadolinium contrast administration (3 min), two dimensional T1-weighted fast-field-echo sequences with an inversion-recovery prepulse will be used. A long inversion time (520 ms) will be used to identify intraventricular thrombus as a LV mass with low-signal intensity surrounded by high-signal intensity structures.
Silent brain infarcts (SBI) | Within 10 days after enrollment
  SBIs diagnosis entails the presence of a focal lesion > 3 mm that meets one of the three following criteria: 1) high signal on DWI isotropic images and low signal on the map of apparent diffusion coefficient (ADC). DWI sequence allows to detecting ischemic lesions (4 hours) and assessing their chronology. (2) cavitary lesion hyperintense on T2, with no signal (or low) in the FLAIR sequence usually surrounded by a ring gliotic hyperintense, hypointense on T1). (3) hyperintense lesion on T2 / T1 hypointense with prior distribution defect known or new in a follow-up study. The studies will be interpreted by a neuroradiologist blinded to clinical and echocardiographic information. For the assessment of whether the brain infarct is clinically silent, a medical history and physical examination focused on neurological symptoms will be performed including for that purpose the National Institute of Health (USA) questionnaire.
Cognitive impact of SBIs | Within 10 days after enrollment
  Cognitive impact of SBIs assessed by MMSE. The Mini Mental State Examination (MMSE) is a tool that can be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30, and the minimum score is 0. A score of 23 or lower is indicative of cognitive impairment.
  The following three cut-off levels are employed to classify the severity of cognitive impairment: no cognitive impairment = 24-30; mild cognitive impairment = 18-23; severe cognitive impairment = 0-17.
Neuropsychiatric impact of SBIs | Within 10 days after enrollment
  Neuropsychiatric impact of SBIs assessed by the Beck Depression Inventory. The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression; each set is ranked in terms of severity and scored from 0 to 3. The maximun score for the whole test is 63 and the lowest is 0. The cut-off scores with patients diagnosed as having an affective disorder are the following: none or minimal depression is < 10; mild to moderate depression is 10-18; moderate to severe depression is 19-29; and severe depression is 30-63.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bermejo Thomas, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hospital General Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bermejo J, Benito Y, Alhama M, Yotti R, Martinez-Legazpi P, Del Villar CP, Perez-David E, Gonzalez-Mansilla A, Santa-Marta C, Barrio A, Fernandez-Aviles F, Del Alamo JC. Intraventricular vortex properties in nonischemic dilated cardiomyopathy. Am J Physiol Heart Circ Physiol. 2014 Mar 1;306(5):H718-29. doi: 10.1152/ajpheart.00697.2013. Epub 2014 Jan 10. PMID 24414062
- [Result] Rossini L, Martinez-Legazpi P, Vu V, Fernandez-Friera L, Perez Del Villar C, Rodriguez-Lopez S, Benito Y, Borja MG, Pastor-Escuredo D, Yotti R, Ledesma-Carbayo MJ, Kahn AM, Ibanez B, Fernandez-Aviles F, May-Newman K, Bermejo J, Del Alamo JC. A clinical method for mapping and quantifying blood stasis in the left ventricle. J Biomech. 2016 Jul 26;49(11):2152-2161. doi: 10.1016/j.jbiomech.2015.11.049. Epub 2015 Nov 30. PMID 26680013
- [Result] Vermeer SE, Longstreth WT Jr, Koudstaal PJ. Silent brain infarcts: a systematic review. Lancet Neurol. 2007 Jul;6(7):611-9. doi: 10.1016/S1474-4422(07)70170-9. PMID 17582361
- [Result] Martinez-Legazpi P, Rossini L, Perez Del Villar C, Benito Y, Devesa-Cordero C, Yotti R, Delgado-Montero A, Gonzalez-Mansilla A, Kahn AM, Fernandez-Aviles F, Del Alamo JC, Bermejo J. Stasis Mapping Using Ultrasound: A Prospective Study in Acute Myocardial Infarction. JACC Cardiovasc Imaging. 2018 Mar;11(3):514-515. doi: 10.1016/j.jcmg.2017.06.012. Epub 2017 Oct 5. No abstract available. PMID 28917683